CLINICAL TRIAL: NCT01768793
Title: Weight Management in Obese Pregnant Underserved African American Women
Acronym: LIFE-Moms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201110073; 5U01DK094416 (NIH)
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Obesity; Pregnancy; Weight Gain
Keywords: Obesity; Pregnancy; Body Weight Changes; Diet Therapy
MeSH Terms: conditions — Obesity; Weight Gain; Body Weight Changes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parents As Teachers + Lifestyle Int. (Experimental): Participants assigned to this group will receive Parents As Teachers Plus (PAT+). This will be a diet and physical activity lifestyle intervention integrated within the standard Parents As Teachers home visiting curriculum. There will be a total of 28 home visits, delivered over 24 months (6 month prenatal phase and 18 month post-partum phase).
  Interventions: Behavioral: Parents As Teachers Plus (PAT+)
- Standard Parents as Teachers (PAT) (Active Comparator): Participants assigned to this group will receive the standard Parents As Teachers (PAT) home visiting curriculum, focusing on parenting and child development. There will be a total of 28 home visits, delivered over 24 months (6 month prenatal phase and 18 month post-partum phase).
  Interventions: Behavioral: Standard Parents As Teachers (PAT)

INTERVENTIONS:
Behavioral: Standard Parents As Teachers (PAT) — Participants will receive visits by Parent Educators, who will deliver the standard PAT curriculum. Participants will receive 28 total visits over the course of approximately 2 years.
  Arms: Standard Parents as Teachers (PAT)
Behavioral: Parents As Teachers Plus (PAT+) — Participants will receive the standard PAT curriculum, plus lifestyle intervention focusing on healthy diet and exercise, through 28 home visits over the course of approximately 2 years.
  Arms: Parents As Teachers + Lifestyle Int.

SUMMARY:
This project will test a novel lifestyle intervention to help overweight and obese socioeconomically disadvantaged African American women achieve healthy weight control during and after pregnancy and improve the health of their offspring. The treatment will be given through an existing national home visiting program, Parents As Teachers (PAT), which will facilitate sustainability and nationwide dissemination, if effective. We hypothesize that compared with standard PAT monitoring and counseling (PAT), women randomized to the lifestyle intervention program (PAT+) will have a lower percentage who exceed Institute of Medicine recommendations for gestational weight gain.

DETAILED DESCRIPTION:
Maternal overweight/obesity and inappropriate gestational weight gain increase both maternal and neonatal morbidity and mortality. In addition, offspring of overweight/obese women are at increased risk for neurodevelopmental delay, becoming obese, and developing metabolic diseases. Women who are socioeconomically disadvantaged (SED), especially from African American populations, are particularly susceptible to adverse pregnancy-related outcomes because of their high prevalence rates of obesity. Therefore, successful weight management during pregnancy in SED, African American women has considerable public health implications. We have experience in testing lifestyle interventions among SED nonpregnant women that have been implemented and sustained within community organizations such as Parents As Teachers (PAT), a national home visiting program that provides parent-child education and services free-of-charge to high-needs women, prenatally and post-partum, with up to 25 home visits per year until kindergarten. We propose to conduct a 24-month (6-month prenatal and 18-month post-partum) randomized, controlled trial in overweight and obese SED African American women to evaluate the ability of an innovative lifestyle intervention program (PAT+), delivered by PAT parent educators during prenatal and post-partum home visits, to improve maternal and neonatal/infant weight, metabolic and health outcomes, relative to the standard PAT program (PAT). A programmatic evaluation will determine the applicability of the PAT+ intervention in real world settings by measuring programmatic reach, implementation, acceptability, and sustainability. If effective, PAT+ can be disseminated through this national organization, which currently reaches over 249,000 mothers and 319,000 children participating in 2,173 PAT programs across all 50 states.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, African American, Socioeconomically disadvantaged
* Established prenatal care at our clinic before 15-6/7 weeks gestation
* Singleton viable pregnancy
* Gestational age 9 to 15 weeks
* Body Mass Index (BMI) of 25-45 kg/m²

Exclusion Criteria:

* Diagnosis of diabetes prior to pregnancy, or test results suggestive of pre-pregnancy diabetes
* Current use of certain medications
* Contraindications to aerobic exercise in pregnancy
* History of contraindicated medical conditions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 267 (Actual)
Dates: Start 2012-10; Primary Completion 2016-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Percent of women whose gestational weight gain exceeds Institute of Medicine recommendations | Delivery (when the baby is delivered)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Cabre HE, Drews KL, Pomeroy J, Keadle SK, Arteaga SS, Franks PW, Haire-Joshu D, Knowler WC, Pi-Sunyer X, Van Horn L, Wing RR, Cahill AG, Clifton RG, Couch KA, Gallager D, Josefson JL, Joshipura K, Klein S, Martin CK, Peaceman AM, Phelan S, Thom EA, Redman LM; LIFE-Moms Research Group. LIFE-Moms: effects of multicomponent lifestyle randomized control trial on physical activity during pregnancy in women with overweight and obesity. Int J Behav Nutr Phys Act. 2025 Sep 30;22(1):119. doi: 10.1186/s12966-025-01805-9. PMID 41029405
- [Derived] Flanagan EW, Drews KL, Cade WT, Franks PW, Gallagher D, Phelan S, Van Horn L, Redman LM. Metabolic Health and Heterogenous Outcomes of Prenatal Interventions: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2528264. doi: 10.1001/jamanetworkopen.2025.28264. PMID 40839263
- [Derived] Mittendorfer B, Patterson BW, Haire-Joshu D, Cahill AG, Cade WT, Stein RI, Klein S. Insulin Sensitivity and beta-Cell Function During Early and Late Pregnancy in Women With and Without Gestational Diabetes Mellitus. Diabetes Care. 2023 Dec 1;46(12):2147-2154. doi: 10.2337/dc22-1894. PMID 37262059
- [Derived] Cade WT, Mittendorfer B, Patterson BW, Haire-Joshu D, Cahill AG, Stein RI, Schechtman KB, Tinius RA, Brown K, Klein S. Effect of excessive gestational weight gain on insulin sensitivity and insulin kinetics in women with overweight/obesity. Obesity (Silver Spring). 2022 Oct;30(10):2014-2022. doi: 10.1002/oby.23533. PMID 36150208
- [Derived] Redman LM, Drews KL, Klein S, Horn LV, Wing RR, Pi-Sunyer X, Evans M, Joshipura K, Arteaga SS, Cahill AG, Clifton RG, Couch KA, Franks PW, Gallagher D, Haire-Joshu D, Martin CK, Peaceman AM, Phelan S, Thom EA, Yanovski SZ, Knowler WC; LIFE-Moms Research Group. Attenuated early pregnancy weight gain by prenatal lifestyle interventions does not prevent gestational diabetes in the LIFE-Moms consortium. Diabetes Res Clin Pract. 2021 Jan;171:108549. doi: 10.1016/j.diabres.2020.108549. Epub 2020 Nov 22. PMID 33238176
- [Derived] Tabak RG, Furtado K, Schwarz CD, Haire-Joshu D. Neighborhood Perceptions Among Pregnant African American Women in St. Louis, Missouri, Before and After the Shooting of Michael Brown. Health Equity. 2020 Aug 19;4(1):353-361. doi: 10.1089/heq.2019.0125. eCollection 2020. PMID 32908956
- [Derived] Haire-Joshu D, Cahill AG, Stein RI, Cade WT, Woolfolk CL, Moley K, Mathur A, Schwarz CD, Schechtman KB, Klein S. Randomized Controlled Trial of Home-Based Lifestyle Therapy on Postpartum Weight in Underserved Women with Overweight or Obesity. Obesity (Silver Spring). 2019 Apr;27(4):535-541. doi: 10.1002/oby.22413. PMID 30900408
- [Derived] Peaceman AM, Clifton RG, Phelan S, Gallagher D, Evans M, Redman LM, Knowler WC, Joshipura K, Haire-Joshu D, Yanovski SZ, Couch KA, Drews KL, Franks PW, Klein S, Martin CK, Pi-Sunyer X, Thom EA, Van Horn L, Wing RR, Cahill AG; LIFE-Moms Research Group. Lifestyle Interventions Limit Gestational Weight Gain in Women with Overweight or Obesity: LIFE-Moms Prospective Meta-Analysis. Obesity (Silver Spring). 2018 Sep;26(9):1396-1404. doi: 10.1002/oby.22250. Epub 2018 Sep 6. PMID 30230252
- [Derived] Lewkowitz AK, Lopez JD, Stein RI, Rhoades JS, Schulz RC, Woolfolk CL, Macones GA, Haire-Joshu D, Cahill AG. Effect of a Home-Based Lifestyle Intervention on Breastfeeding Initiation Among Socioeconomically Disadvantaged African American Women with Overweight or Obesity. Breastfeed Med. 2018 Jul/Aug;13(6):418-425. doi: 10.1089/bfm.2018.0006. Epub 2018 Jun 18. PMID 29912571
- [Derived] Cahill AG, Haire-Joshu D, Cade WT, Stein RI, Woolfolk CL, Moley K, Mathur A, Schechtman K, Klein S. Weight Control Program and Gestational Weight Gain in Disadvantaged Women with Overweight or Obesity: A Randomized Clinical Trial. Obesity (Silver Spring). 2018 Mar;26(3):485-491. doi: 10.1002/oby.22070. PMID 29464907
- [Derived] Clifton RG, Evans M, Cahill AG, Franks PW, Gallagher D, Phelan S, Pomeroy J, Redman LM, Van Horn L; LIFE-Moms Research Group. Design of lifestyle intervention trials to prevent excessive gestational weight gain in women with overweight or obesity. Obesity (Silver Spring). 2016 Feb;24(2):305-13. doi: 10.1002/oby.21330. Epub 2015 Dec 26. PMID 26708836
- See also: Study Consortium website — https://lifemoms.bsc.gwu.edu/